CLINICAL TRIAL: NCT04574258
Title: Contrast-enhanced Ultrasound in Thyroid Tumor by Sonozoid
Brief Title: Prospective Multicenter Study on Clinical Application of Sonozoid in Thyroid Tumor
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Department of Interventional Ultrasound, Chinese PLA General Hospital
Other Study IDs: S2020-300-01-01
Record Dates: First submitted 2020-09-18; First posted 2020-10-05 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Ultrasound
Keywords: Thyroid carcinoma
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — FNA or CNB in thyroid carcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sonazoid as a new generation of ultrasound contrast agent. This study based on the features of Sonazoid specific angiography and high mechanical index, the role of Sonazoid in the differential diagnosis of thyroid benign and malignant tumors was explored.

DETAILED DESCRIPTION:
Sonazoid as a new generation of ultrasound contrast agent, was liver specificity (Kupffer cells), macrophages at the very stable period, Kupffer imaging contrast enhancement effect for more than 1 hour, it is mainly used for focal liver lesions of blood vessels and Kupffer phase of ultrasonic imaging, facilitate early detection of small lesions (< 1 cm). Until now, Sonazoid has been mainly focused on liver focal lesions.

CEUS is an effective imaging method to differentiate thyroid nodules, which can achieve diagnostic accuracy of 84~92.5% based on features of low enhancement, uneven enhancement and circular enhancement. However, studies have shown overlapping findings between CEUS qualitative and quantitative criteria for the evaluation of benign and malignant nodules, limitations in the interpretation of tumor microvascular distribution, and no single indicator has sufficient sensitivity or specificity. Therefore, in the evaluation of thyroid nodules, the existing CEUS interpretation of the results is still limited, the need for a new model.

The existing contrast agents, Sonazoid stability is better, can tolerate relatively high mechanical index and penetration; The size of the microspheres was uniform, with 99.9% less than 7 m, most of which were between 2 and 4 m, and the median diameter of the microspheres was 2.6 m. The imaging was more uniform and clear, and the outstanding advantage was that high-frequency (7-20m) imaging could be realized, which was conducive to the exploration of small superficial lesions in patients. However, studies on Sonazoid in superficial organs such as thyroid were extremely rare.

In addition, Sonazoid microspheres is mononuclear phagocytes specificity contrast agents, main mononuclear phagocyte system including monocytes, connective tissue, lymph nodes and spleen macrophages, kupffer cells of the liver, dust cells of the lung, lymphoid tissue in the crisscross DCS etc. Most researches, both at home and abroad, have confirmed that the expression of Macrophages has long been Associated with the malignancy and lymph node metastasis, but negatively correlated with the prognosis. In thyroid carcinoma, tumor-associated Macrophages was significantly higher than that of benign Tumor and follicular adenoma.

Therefore, based on the features of Sonazoid specific angiography and high mechanical index, the role of Sonazoid in the differential diagnosis of thyroid benign and malignant tumors, the degree of tumor differentiation and the risk assessment of lymph node metastasis was explored.

ELIGIBILITY:
Inclusion Criteria:

* (1) The thyroid nodules were mostly solid or solid.
* (2) Patients with thyroid nodules to be punctured or surgically removed;
* (3) Ability to understand, sign informed consent and agree to participate in the investigator;
* (4) No significant risk of bleeding (platelet ≥50x109/L, prothrombin activity ≥50%)

Exclusion Criteria:

* (1) Patients with a history of neck surgery;
* (2) Women during pregnancy and lactation;
* (3) Ultrasound contrast agent exposure history within 1 month;
* (4) Those who are known to be allergic to ultrasound contrast agents;
* (5) Uncontrolled heart failure.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with thyroid nodule who needs to biopsy or surgical resection;
Sampling Method: Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of contrast-enhanced ultrasound in thyroid tumor by Sonazoid. | 10 months
  Pathology as a gold standard, to evaluate the diagnostic performance (sensitivity, specificity and accuracy) in thyroid tumor by Sonazoid.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiao F, Li JM, Han ZY, Liu FY, Yu J, Xie MX, Zhou P, Liang L, Zhou GM, Che Y, Wang SR, Liu C, Cong ZB, Liang P. Multimodality US versus Thyroid Imaging Reporting and Data System Criteria in Recommending Fine-Needle Aspiration of Thyroid Nodules. Radiology. 2023 Jun;307(5):e221408. doi: 10.1148/radiol.221408. PMID 37367448